CLINICAL TRIAL: NCT06180278
Title: A Long-term, Open-label, Low-interventional Safety Study of Inebilizumab in the Treatment of NMOSD (N-MOmentum LT)
Brief Title: Long-term, Open-label, Safety Study of Inebilizumab in Neuromyelitis Optica Spectrum Disorder (NMOSD)
Acronym: N-MOmentum LT
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HZNP-UPL-401
Expanded Access: NCT06590051 (Available)
Record Dates: First submitted 2023-11-17; First posted 2023-12-22 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Neuromyelitis Optica Spectrum Disorder
Keywords: Immunoglobulins; B-cell count; inebilizumab; Uplizna
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Hematologic Tests; inebilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants with NMOSD exposed to inebilizumab (Other): Participants with NMOSD who previously enrolled in N-MOmentum study, who participated for at least 2 years in the open label phase (OLP) of the study, and participants newly initiating inebilizumab treatment will have hematology, chemistry, B-cell count, serum immunoglobulin (Ig) levels, adverse events, concomitant medications list, NMOSD attacks information, antidrug antibody (ADA) status and titers collected.
  Interventions: Other: Blood tests; Drug: Inebilizumab

INTERVENTIONS:
Other: Blood tests — Participants will have blood tests done at each scheduled visit (approximately every 6 months).
Drug: Inebilizumab — Participants with NMOSD who previously enrolled in N-MOmentum study, who participated for at least 2 years in the open label phase (OLP) of the study, and participants newly initiating inebilizumab treatment at the discretion of their treating physician will have hematology, chemistry, B-cell count, serum immunoglobulin (Ig) levels, adverse events, concomitant medications list, NMOSD attacks information, antidrug antibody (ADA) status and titers collected.
  Other Names: UPLIZNA

SUMMARY:
The purpose of this study is to understand the effects of long-term treatment with inebilizumab on circulating levels of immunoglobulins, B-cell counts, and other safety measures, and to further monitor repletion of immunoglobins and B-cell counts in participants with NMOSD who discontinue treatment. The objectives include:

1. To establish the nadir in circulating immunoglobulins (Ig) during chronic treatment with inebilizumab and ascertain the time needed to ensure restoration of pre-treatment baseline serum levels of IgG and IgM after discontinuation of treatment
2. To characterize B-cell counts throughout treatment with inebilizumab and after discontinuation until repletion of Immunoglobulin (Ig levels)
3. To assess long-term safety of inebilizumab
4. To assess other long-term effects of inebilizumab

DETAILED DESCRIPTION:
This study aims to enroll 30 participants who either participated in the open-label period (OLP) of the N-MOmentum study (CD-IA-MEDI-551-1155; NCT02200770), a global registrational study that determined the safety and efficacy of inebilizumab for treatment of NMOSD, or who are newly initiating inebilizumab treatment at the discretion of their physician at participating sites.

Acquired from Horizon in 2024.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or above, and able to provide written informed consent and any locally required authorization (e.g., Health Insurance Portability and Accountability Act [HIPAA] in the United States of America (USA), European Union [EU] Data Privacy Directive in the EU) obtained from the subject/legal representative prior to performing any protocol-related procedures, including screening evaluations.
2. Have completed at least 2 years in the open-label period of the N-MOmentum study or are newly initiating inebilizumab treatment at a participating site.
3. Females of childbearing potential who are sexually active with a nonsterilized male partner must use a highly effective method of contraception as outlined in the protocol (subjects in the Czech Republic only must use 1 additional method of contraception) from screening, and must agree to continue using such precautions for 6 months after treatment with inebilizumab; cessation of contraception after this point should be discussed with a responsible physician.
4. Nonsterilized males who are sexually active with a female partner of childbearing potential must use a male condom plus spermicide (subjects in the Czech Republic only must use 1 additional method of contraception) from Day 1 for 3 months after receipt of last treatment with inebilizumab.
5. Sterilized males, without the appropriate post-vasectomy documentation on the absence of sperm in the ejaculate, who are sexually active with a female partner of childbearing potential must use a condom and spermicide from Day 1 for 3 months after receipt of the last treatment with inebilizumab.

Exclusion Criteria:

1. Have any condition that would place the participant at unacceptable risk of complications, interfere with evaluation of inebilizumab or confound the interpretation of participant safety or study results.
2. Received rituximab or any other B-cell depleting agent after exit from N-MOmentum study, or within the last 12 months prior to screening for non N-MOmentum participants.
3. Known history of allergy or reaction to any component of inebilizumab formulation or history of anaphylaxis following any biologic therapy
4. Have a severe clinically significant infection, including active chronic infection such as hepatitis B
5. Have active or untreated latent tuberculosis
6. Have a history of progressive multifocal leukoencephalopathy (PML)
7. Is severely immunocompromised state
8. Have active malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2028-06-26 (Estimated); Study Completion 2028-06-26 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in serum Ig levels (total Ig, IgG, IgM, IgA, IgE) over time | Up to 42 months
  This will be assessed via serum samples, drawn at the site and processed at a central laboratory, and analyses performed to assess change from baseline over time, as measured by each parameter in mg/dL
Change from baseline in peripheral CD20+ B-cell counts over time | Up to 42 months
  This will be assessed via serum samples, drawn at the site and processed at a central laboratory, and analyses performed to assess change from baseline over time, as measured by each parameter in cells/mL

SECONDARY OUTCOMES:
Change from baseline in hematology over time | Up to 42 months
  The lab parameters being assessed as part of the hematology analyses include the following: platelet count, red blood cell count, other indices of red blood cells, including MCV (mean corpuscle volume), MCH (mean corpuscle hemoglobin), % reticulocyte count, and morphology (shape); white blood count with differential, including neutrophil count, Lymphocyte count, monocyte count, eosinophils, and basophils; hemoglobin and hematocrit.
Change from baseline in clinical chemistry over time | Up to 42 months
  The lab parameters being assessed as part of clinical chemistry include blood urea nitrogen (BUN), creatinine, aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase.
Incidence of serious infections | Up to 42 months
Incidence of viral reactivation | Up to 42 months
Incidence of progressive multifocal leukoencephalopathy (PML) | Up to 42 months
Incidence of other opportunistic infections | Up to 42 months
Incidence of malignancies | Up to 42 months
Incidence of infusion reactions | Up to 42 months
Number of protocol-defined NMOSD attacks | Up to 42 months
Percentage of protocol-defined NMOSD attacks | Up to 42 months
Incidence of Anti-drug antibody (ADA) directed against Inebilizumab status and titers | Up to 42 months

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (11):
- United States (2):
  - Wayne State University School of Medicine, Detroit, Michigan
  - Baylor College of Medicine, Houston, Texas
- Prince of Wales Hospital (PWH) - The Chinese University of Hong Kong (CUHK) - Ophtalmology, Hong Kong, China
- Vseobecna fakultni nemocnice v Praze - Neurologicka klinika, Prague, Czechia
- Szegedi TudomÃ¡nyegyetem, Ã OK, Szent-GyÃ¶rgyi Albert Klinikai KÃ¶zpont - NeurolÃ³giai OsztÃ¡ly, Szeged, Csongrád megye, Hungary
- Poland (2):
  - Uniwersyteckie Centrum Kliniczne WUM - Oddzial Kliniczny Neurologii, Warsaw, Masovian Voivodeship
  - M.A.-Lek A.M. Maciejowscy S.C. Centrum Terapii SM, Katowice, Silesian Voivodeship
- South Korea (3):
  - National Cancer Center - Neurology Clinic, Goyang-si, Gyeonggido [Kyonggi-do]
  - Seoul National University Hospital, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp
  - Samsung Medical Center - Pediatric Neurology, Seoul, Seoul Teugbyeolsi [Seoul-T'ukp
- Khon Kaen University, Srinagarind Hospital - Division of Neurology, Depart, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com